CLINICAL TRIAL: NCT02158156
Title: Effect of Aerobic Training in Patients With Oculopharyngeal Muscular Dystrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Karen Brorup Heje Pedersen, Bsc Medicine, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H2-2013-066(A)
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Oculopharyngeal Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Excercise (Experimental): 10 weeks of home training on a cycle-ergometer. Exercise 30 minutes every other day or at least three times a week.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Ten weeks of home-training on a cycle ergometer 3 times a week for 30 minutes.

SUMMARY:
The investigators want to investigate if patients with Oculopharyngeal Muscular Dystrophy can improve fitness by home-training on a cycle ergometer 30 minute, 3 times a week for 10 weeks.

Participants will be evaluated on maximal oxygen consumption and maximal workload measured by an incremental test at baseline and at the end of the exercise period.

ELIGIBILITY:
Inclusion Criteria:

* Danish patients with Oculopharyngeal muscular dystrophy

Exclusion Criteria:

* Patients who are too week to train on an cycle-ergometer for 10 weeks
* Patients with other health issues wich confound the interpretation of the efficacy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy based on VO2max | 10 weeks
  Difference in VO2max measured before and after intervention

SECONDARY OUTCOMES:
SF-36 Questionaire | 10 weeks
  Changes in self-rated health from baseline to end of intervention
6 minute walk test | 10 weeks
  Changes in walking distance from baseline to end of intervention
Intensity in maximal load (Watt) | 10 weeks
  Changes in maximal load (watt) in the VO2max-test from baseline to end of intervention.
Level of plasma creatine kinase | 10 weeks
  Marker for exercise-induced muscle damage. Taken week 0,3 and 10.
Level of plasma myoglobin | 10 weeks
  Marker for excercise-induced muscle damage, taken week 0, 3 and 10.
6 minute walk test | 10 weeks
  Changes in walking distance in the test from baseline to end of intervention.
A five-time-repetition-sit-to-stand-test | 10 weeks
  Changes in time of five repetitions from baseline to end of intervention
A 14-step-stair-test | 10 weeks
  Changes in time completing the test from baseline to end of intervention
Dynamometry | 10 weeks
  Changes in external force production from baseline to end of intervention. Dynamometry are measured on hip flexion, dorsal foot flexion, plantar foot flexion, knee flexion, knee extension, and elbow flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Karen BH Pedersen, Bsc.med., Principal Investigator — Neuromuscular Research Unit, Rigshospitalet, Denmark
Locations (1):
- Neuromuscular Research Unit, Copenhagen, Denmark

REFERENCES:
- See also: Website of the Neuromuscular Research Unit, Rigshospitalet, Copenhagen, Denmark — http://www.neuromuscular.dk